CLINICAL TRIAL: NCT05306834
Title: Stopping Cognitive Decline and Dementia by Fighting Covert Cerebral Small Vessel Disease
Acronym: SHIVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2021/22
Record Dates: First submitted 2022-02-25; First posted 2022-04-01 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Small Vessel Diseases; Stroke; Dementia
Keywords: Cognitive decline; Dementia; Stroke; Small vessel disease; Healthy brain aging; Brain imaging; Adaptive optics; Optical coherence tomography angiography; Prevention; Risk prediction; Genomic; Multiomics; Proteomics; Metabolomics
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Stroke; Dementia; Cognitive Dysfunction | interventions — Blood Specimen Collection; Neuroimaging; Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal cSVD patient group (Active Comparator): little or no white matter hyperintensities
  Interventions: Procedure: Retinal Imaging; Genetic: Blood sample; Procedure: Evaluation of cardiovascular risks; Procedure: Brain imaging (MRI); Other: Cognitive Tests; Other: Geriatric Depression Scale (GDS); Other: Instrumental Activities of Daily Living (IADL); Diagnostic Test: Unipodal standing test; Other: Walking speed measurement
- Extensive cSVD patient group (Active Comparator): moderate to severe white matter hyperintensities
  Interventions: Procedure: Retinal Imaging; Genetic: Blood sample; Procedure: Evaluation of cardiovascular risks; Procedure: Brain imaging (MRI); Other: Cognitive Tests; Other: Geriatric Depression Scale (GDS); Other: Instrumental Activities of Daily Living (IADL); Diagnostic Test: Unipodal standing test; Other: Walking speed measurement

INTERVENTIONS:
Procedure: Retinal Imaging — Auto-Refractometry / Adaptative Optics (OA) / Swept Source Optical Coherence Tomography (SS-OCT-A) / Globe Axial length measurements / Color Retinophotography of the retina.
Genetic: Blood sample — Analyses of molecular biomarkers including
Procedure: Evaluation of cardiovascular risks — Measurement of blood pressure and arterial stiffness
Procedure: Brain imaging (MRI) — 3DT1 / 3DFLAIR / T2GRE / DTI 15 directions (and B0MAP)
Other: Cognitive Tests — Mini Mental State Examination (MMSE) / Montreal Cognitive Assessment (MoCA) / 16 items Free and Cued Recall (RL/RI 16 items) / Trail Making Test A et B (TMT A et B) / Frontal Assessment Battery (FAB) / Phonemic (letter P) and semantic (animals) verbal fluency tests / Digit Symbol Substitution Test (DSST)
Other: Geriatric Depression Scale (GDS) — 15 items
Other: Instrumental Activities of Daily Living (IADL) — Instrumental Activities of Daily Living (IADL)
Diagnostic Test: Unipodal standing test — Unipodal standing test
Other: Walking speed measurement — over 5 meters

SUMMARY:
Cerebral small Vessel Disease (cSVD), characterized by an alteration of the structure and function of small penetrating brain arteries, is highly prevalent in older persons from the general population and represents a leading cause of stroke and a major contributor to cognitive decline and dementia risk. In France >4 million persons aged 60+ are estimated to have moderate to extensive covert cSVD (ccSVD), i.e. features of SVD on brain imaging without a history of clinical stroke. Better detection and management of covert cSVD would have a major impact on preventing disability and costs related to stroke, cognitive impairment and dementia. However, there are no specific mechanistic treatments for cSVD and hardly any recommendations worldwide on how to prevent and treat cSVD and related cognitive impairment. The aim of the present study, through the identification of novel cutting-edge multimodal biomarkers, is to develop innovative diagnostic and risk prediction tools for cSVD and its complications and to contribute to accelerating the discovery of novel drug targets and therapeutics strategies for cSVD.

DETAILED DESCRIPTION:
cSVD is by far the most prevalent vascular contributor to cognitive impairment in the population. However, accurate quantitative estimates of the predictive ability of cSVD for dementia risk are lacking. Moreover, stratification of cognitive decline and dementia risk in cSVD patients according to imaging characteristics as well as evidence of coexisting neurodegenerative disease and vascular comorbidity are lacking. Hypertension is the strongest known risk factor for cSVD but there are currently no guidelines for the management of cSVD (or emerging guidelines based on weak evidence, and no specific mechanism-based treatments, leading to empirical and heterogeneous clinical practice, which in most instances consists of ignoring these lesions. This clinical blind spot represents a major "missed opportunity" for the prevention of cognitive decline and dementia.

This study aims to explore the relation of brain and retinal microvasculature image characteristics (imaging biomarkers), as well as molecular biomarkers derived from blood, with presence or absence of extensive cSVD and with cognitive and other clinical characteristics in two groups of 200 patients 60+ years of age. The first group will consist of patients with little or no white matter hyperintensities on brain MRI (no or minor MRI features of cSVD); while the second will include patients with moderate to severe white matter hyperintensities (MRI features of extensive cSVD).

This will create a unique deeply characterized resource for epidemiological and mechanistic investigations of cSVD, which can also serve as a pilot setting to test the trajectories and requirements for individualized patient care of cSVD patients.

The combination of retinal microvascular measurements using innovative multimodal imaging is entirely novel to our knowledge. In the context of the RHU SHIVA program, the same retained imaging protocol will be implemented for 400 young adults, which will provide insight into trajectories of these retinal biomarkers across the adult lifespan).

For the molecular biomarkers allow the validation of genomic, epigenomic, transcriptomic, proteomic, and metabolomic biomarkers for cSVD identified through secondary use of large existing cohort studies in the general population (3C, i-Share cohorts), in persons with memory complaints (MEMENTO cohort), and in collaboration with other cohorts with the Cohorts for Heart and Aging Research in Genomic Epidemiology (CHARGE) consortium, also as part of the RHU SHIVA program.

ELIGIBILITY:
Inclusion Criteria:

For the extensive cSVD patient group

1. For the extensive cSVD patient group included in the LEOPOLD trial:

   * Patients aged 60 to 88 years,
   * Patients included in the LEOPOLD trial and having performed their brain MRI on SIEMENS PRISMA machine
   * Being affiliated or beneficiary of the French national health insurance ("sécurité sociale"),
   * Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research study).
2. For the extensive cSVD patient group not included in the LEOPOLD trial:

   * Patients aged 60 to 88 years,
   * Patients with a cognitive complaint MMSE ≥ 20 performed in the 6 months before inclusion, associated or not with impaired cognitive tests and/or diaognosis of incipient dementia without pronounced cognitive deterioration,
   * Patients with a socio-educational level ≥ 3,
   * Patients with a moderate to high grade of hypersignals on an MRI OR on an CT scan performed prior inclusion (grades C and D of the modified Scheltens scale or grade 2/3 Fazekas),
   * Arterial hypertension defined by a Systolic Blood Pressure (SBP) and / or Diastolic Blood Pressure (DBP) ≥ 140/90 mmHg (according to the definition of the national health authority [HAS]), treated or not, confirmed within the previous 12 months or at the latest on the day of inclusion.
   * Being affiliated or beneficiary of the French national health insurance ("sécurité sociale"),
   * Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research study)

For the minimal cSVD patient group:

* Patients aged 60 to 88 years,
* Patients with a cognitive complaint (MMSE ≥ 20 performed at the SHIVA inclusion visit or in the 6 monts prior the visit) associated or not with impaired cognitive tests and/or diagnosis of incipient dementia without pronounced cognitive deterioration,
* Patients with little or no white matter hypertensities on brain MRI (grades 0 or 1 on the Fazekas scale); without lacunes or microbleeds,
* Arterial hypertension defined by a Systolic Blood Pressure (SBP) and / or Diastolic Blood Pressure (DBP) ≥ 140/90 mmHg (according to the definition of the national health authority [HAS]), treated or not, confirmed within the previous 12 months or at the latest on the day of inclusion. Blood pressure values for this inclusion criterion can be objectified by several self-measurements performed by the patient at home for 3 days in a sitting or lying position (3 measurements on sitting or lying position and 3 measurements in standing position).
* Being affiliated or beneficiary of the French national health insurance ("sécurité sociale"),
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research study

Exclusion Criteria:

For Extensive cSVD patient group :

1. For the extensive cSVD patient group also included in the LEOPOLD trial:

   * patients with severe myopia greater than -6 dioptres
   * partients with known allergy to Tropicamide (Mydriaticum®)
   * patients with an extensive cataract
   * patients with ptosis
2. For the extensive cSVD patient group not included in the LEOPOLD trial:

   * Orthostatic hypotension defined by a decrease of 20 mmHg in SBP and / or 10 mmHg in DBP in a standing position at 3 minutes sought in the previous 3 months or on the day of inclusion,
   * Very severe renal impairment (creatinine clearance less than 15 ml / min) on a blood test dating back less than one year,
   * Secondary hypertension: renovascular hypertension, primary hyperaldosteronism, pheochromocytoma...
   * Contraindication to MRI (presence of a ferromagnetic foreign body, in particular certain intracranial clips, certain heart valves, an intraocular foreign body, metal prosthesis, subject carrying a pacemaker, subject carrying prosthetic heart valves incompatible with MRI. ventricular shunt, claustrophobia),
   * Associated severe diseases, with a life expectancy of less than 3 months,
   * Physical problems likely to interfere with the feasibility of the tests (sight, hearing, etc.),
   * Existence of dementia of which the etiology is distinct from Alzheimer's disease, vascular or mixed dementia
   * Persons under tutorship or curatorship,
   * Patients with loss of autonomy living in EHPAD (nursing home)
   * patients with severe myopia greater than -6 dioptres
   * participants with known allergy to Tropicamide (Mydriaticum®)
   * patients with an extensive cataract
   * patients with ptosis

For the minimal cSVD patient group:

* Orthostatic hypotension defined by a decrease of 20 mmHg in SBP and / or 10 mmHg in DBP in a standing position at 3 minutes sought in the previous 3 months or on the day of inclusion,
* Very severe renal impairment (creatinine clearance less than 15 ml / min) on a blood test dating back less than one year,
* Secondary hypertension: renovascular hypertension, primary hyperaldosteronism, pheochromocytoma...
* Contraindication to MRI (presence of a ferromagnetic foreign body, in particular certain intracranial clips, certain heart valves, an intraocular foreign body, metal prosthesis, subject carrying a pacemaker, subject carrying prosthetic heart valves incompatible with MRI. ventricular shunt, claustrophobia),
* Associated severe diseases, with a life expectancy of less than 3 months,
* Physical problems likely to interfere with the feasibility of the tests (sight, hearing, etc.),
* Existence of dementia of which the etiology is distinct from Alzheimer's disease, vascular or mixed dementia
* Persons under tutorship or curatorship,
* Patients with loss of autonomy living in EHPAD (nursing home)
* Patients with severe myopia greater than -6 dioptries
* Patients with known allergy to Tropicamide (Mydriaticum®)
* Patients with an extensive cataract
* Patients with ptosis

Ages: 60 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of images and the molecular data | Day 0 and Year 3
  This comparison should help identify relevant biomarkers to characterize and categorize cSVD. We will also more broadly look at the association of retinal microvascular markers and molecular biomarkers with all available MRI-markers of cSVD (beyond the presence or absence of extensive white matter hyperintensities that defines the cases and controls).

SECONDARY OUTCOMES:
Degree of association between retinal and brain marker | Day 0, Year 1 and Year 3
  Degree of association between retinal and brain marker
Degree of association between brain, microvascular and retinal marker | Day 0, Year 1, Year 2 and Year 3
  Data relating to cardiovascular risk factors / clinic data / the results of the cognitive tests, /the results of pan-genomic genotypes obtained by pan-genome genotyping or sequencing (and from blood samples) and other molecular markers
Correlation between retinal micovascular biomarkers | Day 0, Year 1, Year 2 and Year 3
  SS-OCT-A (swept source optical coherence tomography angiography) and OA(Adaptive Optic)
Reproducibility and time course of retinal vascular biomarkers | Between Day 0 and Year 1
  SS-OCT-A (swept source optical coherence tomography angiography) and OA (Adaptive Optic)
Detecting, classifying and quantifying markers of retinal microvascular lesions | up to year 3
  Performance image acquisition -OCT-A (swept source optical coherence tomography angiography) and OA (Adaptive Optic)
Comparison of the results in the Shiva study and SHIVA share study | through study completion, an average of 3 year
  Comparison of the association results and mean distributions observed in SHIVA with those observed in the SHIVA-Share
Occurrence of incident stroke, dementia and death during follow-up. | through study completion, an average of 3 year
  Association of all imaging or molecular biomarkers with the occurrence of incident stroke, dementia and death during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HANON, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marc JOLIOT, Dr, Study Chair — Unité CNRS UMR5296, Groupe d'Imagerie; Cécile DELCOURT, Dr, Study Chair — Centre INSERM U1219 Bordeaux Population Health
Locations (2):
- France (2):
  - Bordeaux Hospital, Bordeaux
  - Broca Hospital, Paris

IPD SHARING:
Plan to Share IPD: No